CLINICAL TRIAL: NCT05789082
Title: A Phase Ib/II, Open-Label, Multicenter Study Evaluating the Safety, Activity, and Pharmacokinetics of Divarasib as a Single Agent or in Combination With Other Anti-Cancer Therapies in Patients With Previously Untreated Advanced Or Metastatic Non-Small Cell Lung Cancer With a KRAS G12C Mutation
Brief Title: A Study Evaluating the Safety, Activity, and Pharmacokinetics of Divarasib as a Single Agent or in Combination With Other Anti-Cancer Therapies in Participants With Previously Untreated Advanced or Metastatic Non-Small Cell Lung Cancer With a KRAS G12C Mutation
Acronym: KRAScendo 170
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO44426; 2022-003048-28 (EudraCT Number); 2023-507171-22-00 (EU CTIS Number)
Record Dates: First submitted 2023-02-21; First posted 2023-03-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Cisplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Cohorts B, C, D, and a subset of Cohort A follow non-randomized allocation; other subsets of Cohort A are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A - Combination Dose Finding + Dose Expansion (Experimental): Participants will be enrolled in different cohorts to receive divarasib (different dose levels will be evaluated) once a day (QD) combined with pembrolizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W).
  During the expansion stage, some participants are planned to be randomized to one divarasib combination dose level; other participants are planned to be randomized to another divarasib combination dose level. Divarasib will be given in combination with pembrolizumab.
  Interventions: Drug: Divarasib; Drug: Pembrolizumab
- Cohort B - Combination Dose Finding + Dose Expansion (Experimental): Participants enrolled in this cohort will receive divarasib (different dose levels will be evaluated) QD combined with pembrolizumab 200 mg IV Q3W plus investigator's choice of platinum-based chemotherapy (carboplatin or cisplatin) and pemetrexed.
  Interventions: Drug: Divarasib; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed
- Cohort C - Dose Expansion (Experimental): Participants enrolled in this cohort will receive one dose level of divarasib QD.
  Interventions: Drug: Divarasib
- Cohort D - Dose Expansion (Experimental): Participants enrolled in this cohort will receive one dose level of divarasib QD.
  Interventions: Drug: Divarasib

INTERVENTIONS:
Drug: Divarasib — Participants will receive divarasib orally (PO), QD on days 1-21 of each 21-day cycle.
Drug: Pembrolizumab — Participants will receive a 200 mg IV infusion of pembrolizumab Q3W on Day 1 of each 21-day cycle.
  Arms: Cohort A - Combination Dose Finding + Dose Expansion; Cohort B - Combination Dose Finding + Dose Expansion
Drug: Carboplatin — Participants will receive IV carboplatin Q3W for four 21-day cycles.
  Arms: Cohort B - Combination Dose Finding + Dose Expansion
Drug: Cisplatin — Participants will receive IV cisplatin Q3W for four 21-day cycles.
  Arms: Cohort B - Combination Dose Finding + Dose Expansion
Drug: Pemetrexed — Participants will receive IV pemetrexed Q3W.
  Arms: Cohort B - Combination Dose Finding + Dose Expansion

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), and activity of single-agent divarasib or combined with other anti-cancer therapies in participants with previously untreated, advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of Biomarker eligibility
* Pre-treatment tumor tissue along with an associated pathology report is required for all participants enrolled on study. Representative tumor specimens must be in formalin-fixed, paraffin embedded (FFPE) blocks (preferred) or 15 unstained, freshly cut, serial slides. Although 15 slides are required, if only 10 slides are available, the participant may be eligible for the study following consultation with the Sponsor.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Histologically or cytologically documented locally advanced unresectable or metastatic NSCLC that is not eligible for curative surgery and/or definitive chemoradiotherapy
* No prior systemic treatment for advanced unresectable or metastatic NSCLC
* Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Additionally, for participants in cohort D, measurable brain metastases defined as at least 5 millimeters and twice the slice thickness, but less than 20 mm, that is asymptomatic and does not require local therapy at the time of enrollment.

Exclusion Criteria:

* Known concomitant second oncogenic driver with available targeted treatment
* Squamous cell histology NSCLC
* Symptomatic, untreated, or actively progressing CNS metastases (Cohorts A, B, and C)
* Prior treatment with a KRAS G12C inhibitor
* Known hypersensitivity to any of the components of divarasib or pembrolizumab; or known hypersensitivity to pemetrexed, carboplatin, or cisplatin (Cohort B only)
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis, active tuberculosis, significant cardiovascular disease within 3 months prior to initiation of study treatment
* History of malignancy other than NSCLC within 5 years prior to initiation of study treatment, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate more >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal breast carcinoma in situ, or Stage I uterine cancer
* Uncontrolled tumor related pain, pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures, uncontrolled or symptomatic hypercalcemia
* Co-morbid condition that is an absolute contraindication to treatment with corticosteroids
* Inability or unwillingness to take prophylactic treatments such as corticosteroids, anti-emetics, folic acid, or vitamin B12 supplementation.
* Participants with brain metastases for whom complete surgical resections is clinically appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2032-01-29 (Estimated); Study Completion 2032-01-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Baseline until 60 days after the final dose of study treatment or until initiation of another anti-cancer therapy, whichever occurs first (up to approximately 5 years)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 5 years
  The percentage of participants who experience a complete response or partial response, as determined by the investigator, according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of Response (DOR) | Approximately 5 years
  The time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Progression Free Survival (PFS) | Approximately 5 years
  The time from randomization, or date of first treatment for participants enrolled prior to the expansion stage, to the first occurrence of disease progression or death from any cause during the study (whichever occurs first), as determined by the investigator according to RECIST v1.1
Number of Participants Reporting Presence, Frequency, Severity, and/or Degree of Interference with Daily Function of Symptomatic Side Effects as Assessed Through the Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Approximately 5 years
Change from Baseline in Symptomatic Side Effects, as Assessed Through use of the PRO-CTCAE | Baseline up to approximately 5 years
Percentage of Participants Reporting "Frequent" or "Almost Constant" Diarrhea During the First Three Cycles of Treatment According to the PRO-CTCAE Criteria | Approximately 5 years
Percentage of Participants Reporting "Severe" or "Very Severe" Nausea or Vomiting During the First Three Cycles of Treatment According to the PRO-CTCAE | Approximately 5 years
Frequency of Participant's Response of the Degree they are Troubled with Treatment Symptoms, as Assessed Through use of the Single-item European Organisation for Research and Treatment of Cancer (EORTC) Item List 46 (IL46) | Approximately 5 years
Plasma or CSF Concentration of Divarasib at Specified Timepoints | Approximately 5 years
  Optional CSF samples may be collected at the time of disease progression or at any time during the study for participants who have provided written consent and if collection of CSF sample is deemed clinically feasible. Matched optional plasma samples may be drawn at the same time.
Identification of Divarasib Recommended Dose | Approximately 5 years
  The recommended dose will be based upon the totality of safety, activity, and PK data.
Central Nervous System (CNS) Response | Approximately 5 years
  Defined as the percentage of participants who experience a complete response or partial response in the brain, as determined by the investigator according to modified RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (70):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - City of Hope - Seacliff, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UCSD Moores Cancer Center, La Jolla, California
  - City of Hope - Long Beach Elm, Long Beach, California
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists - SOUTH - SCRI - PPDS, Fort Myers, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, St. Petersburg, Florida
  - Florida Cancer Specialists - EAST - SCRI - PPDS, West Palm Beach, Florida
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Cancer Center, New York, New York
  - Mount SInai Medical Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc, Blacksburg, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Argentina (3):
  - Hospital Britanico, Buenos Aires
  - Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - Clinique Ste-Elisabeth, Namur
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (2):
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (3):
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- China (3):
  - Hunan Cancer Hospital, Changsha
  - Harbin Medical University Cancer Hospital, Harbin
  - Shanghai Pulmonary Hospital, Shanghai
- Israel (3):
  - Rambam Medical Center, Haifa
  - Rabin MC, Petah Tikva
  - Tel Aviv Sourasky Medical Ctr, Tel Aviv
- Italy (4):
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - A.O. Universitaria S. Luigi Gonzaga, Orbassano, Piedmont
- Japan (5):
  - National Cancer Center Hospital East, Chiba
  - Kindai University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Netherlands (2):
  - NKI The Netherlands Cancer Institute, Amsterdam
  - UMC St Radboud, Nijmegen
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Krakowski Szpital Specjalistyczny im sw. Jana Paw?a II, Krakow
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - ICO Badalona-H.U. Germans Trias i Pujol, Badalona, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan Uni Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- United Kingdom (2):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Barts & London School of Med, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing